CLINICAL TRIAL: NCT04586946
Title: An Observational Study of the Effects of Nocturnal Hypoxaemia on Patients With Fibrotic Interstitial Lung Disease
Brief Title: FIBRotic Interstitial Lung Disease and Nocturnal OXygen
Acronym: FIBRINOX
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Fibrinox 1.0
Record Dates: First submitted 2018-12-17; First posted 2020-10-14 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2020-10

CONDITIONS: Idiopathic Pulmonary Fibrosis; Obstructive Sleep Apnea; Sleep Disturbance; Sleep Hypoventilation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Sleep Apnea, Obstructive; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted and used to genotype common variants known to be associated with pulmonary fibrosis, including but not limited to Muc5b, TOLLIP and TERT. Serum and plasma will be analysed for solu-ble biomarkers including but not limited to KL-6, SP-A, SP-D, Fas, MMP1, MMP7, clusterin, dynamin, VEGF, CCL18, osteopontin, thrombospondin and inflammatory cytokines. Levels in biomarkers and geno-type frequency will be compared between subgroups of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Home sleep studies - which allow the measurement of breathing while the person sleeps - will be performed on patients with fibrotic interstitial lung disease attending two of the UK's largest respiratory medicine services.The study will investigate at how symptoms, and breathing and exercise tests differ between these two groups after 12 months of study.

DETAILED DESCRIPTION:
The interstitial lung diseases are a group of diseases in which patients develop uncontrolled scarring (called fibrosis) within the lung. This causes failure of the lung and patients become progressively more breathless over time. The commonest of these diseases is idiopathic pulmonary fibrosis and this is a devastating condition with a survival of 3-5 years.

Many people with fibrotic interstitial lung diseases have disrupted sleep as well as low oxygen levels at night or obstructive sleep apnoea (OSA - pauses in breathing at night time due to obstruction of the upper airway).

Patients with low oxygen levels at night have a worse quality of life, with fatigue during the day and survive for less long.

102 patients from specialist clinics at Guy's and St Thomas' and the Royal Brompton and Harefield NHS Foundation Trusts will be recruited. This research is funded by a grant from the British Lung Foundation. The investigators aim to compare patients with and without low oxygen levels at night by observing how their disease and quality of life changes over a year.

Patients will be asked to complete a two-night home sleep study which will involve wearing a probe over the finger connected to a sensor on the wrist. Patients will also be provided with a home spirometer to measure their breathing at home daily during the study.

Lung function testing (which is part of normal clinical practice), a six-minute walk test and quality of life questionnaires will be performed at the beginning of the study. These investigations will be repeated at six and twelve months and this will tell us how night time oxygen levels affect the progression of the disease, quality of life, exercise tolerance, hospitalisation frequency and survival of these patients.

ELIGIBILITY:
Inclusion Criteria:

* MDT diagnosis of fibrotic interstitial lung disease including but not limited to idiopathic pulmonary fibrosis (IPF), non-specific interstitial pneumonitis (NSIP), chronic hypersensitivity pneumonitis (CHP), fibrotic organising pneumonia and unclassifiable fibrotic lung disease.
* Competent to provide written consent in English

Exclusion Criteria:

* Presence of an underlying connective tissue disease
* Daytime/resting hypoxaemia with pO2 <8.0
* Other indication for oxygen therapy
* 3% ODI >15 events/hour studied or established on CPAP
* Predominant emphysema on CT
* Inability to provide informed consent or complete health-related quality of life questionnaires in English
* Current participation in a research project which might alter lung function or sleep study results

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with fibrotic interstitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Quality of life measured by King's Brief Interstitial Lung Disease Questionnaire (K-BILD) | 0 months,12 months
  Change in K-BILD score from baseline at 12 months in patients with nocturnal hypoxaemia vs those without (defined as time spent with SpO2<90% of > 10% total sleep time)

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | 12 months
  Annualised decline in FVC in patients with nocturnal hypoxaemia vs those without
Diffusion capacity of the lung for carbon monoxide (DLCO) | 12 months
  Change in DLCO from baseline at 6 and 12 months in patients with nocturnal hypoxaemia vs those without
Pittsburgh Sleep Quality Index (PSQI) | 0 months, 6 months, 12 months
  PSQI score at baseline, and change at 6 and 12 months in patients with nocturnal hypoxaemia vs those without
Insomnia Severity Index (ISI) | 0 months, 6 months, 12 months
  ISI score at baseline, and change at 6 and 12 months in patients with nocturnal hypoxaemia vs those without
Six-minute walk test (6MWT) | 0 months 6 months, 12 months
  Total distance (in metres) and minimum oxygen saturation during 6MWT at baseline, 6 and 12 months
Exacerbation frequency and hospitalisation | 12 months
  Exacerbation frequency and hospitalisation
Mortality | 12 months
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Alex West, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No
Data will be collected on paper worksheets filed in the site file and web-based electronic clinical record forms provided by Castor EDC, a secure web database which is compliant with GCP regulations, Annex 11 and 21 CFR part 11. It also complies with EU GDPR. All communication to servers is encrypted using TLS (1.1 or 1.2) through HSTS.